CLINICAL TRIAL: NCT03824262
Title: The Comparison of Warming Techniques in Patients Undergoing Open Abdominal Surgery in Litotomy Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Filiz Uzumcugil, Principal Investigator, MD, Asist. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E.308215
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): HICO-VARIOTHERM 550 and Mistral-Air Plus forced-air warming device
  Interventions: Device: HICO-VARIOTHERM 550; Device: Mistral-Air Plus forced air warming device
- Group II (Active Comparator): Mistral-Air Plus forced-air warming device
  Interventions: Device: Mistral-Air Plus forced air warming device

INTERVENTIONS:
Device: HICO-VARIOTHERM 550 — Warming during perioperative period.
  Arms: Group I
Device: Mistral-Air Plus forced air warming device — Warming during perioperative period.

SUMMARY:
The patients scheduled to undergo major abdominal surgery in litotomy position will be randomized into two groups in order to compare the effects of two warming techniques during the intraoperative period.

DETAILED DESCRIPTION:
The patients will be randomized into two groups. All patients will receive prewarming with forced-air warming device for 30 minutes. All patients will receive warmed fluids during intraoperative period. One group will receive warming with only forced-air warming device and the other group will receive warming with both forced-air warming device and water mattress. Timpanic, esophageal and peripheral temperature monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery in litotomy position
* ASA I-II
* Anticipated operation time over 1 hour

Exclusion Criteria:

* Sepsis
* Hypothermia
* Hyperthermia
* Malignant Hyperthermia
* Tyroid dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Body temperature-esophageal probe | Perioperative period-every 15 minutes
  Esophageal probe used to measure core body temperature

SECONDARY OUTCOMES:
Body temperature-tympanic thermometer | Perioperative period-every 15 minutes
  Tympanic thermometer used to measure body temperature
Body temperature-skin thermometer | Perioperative period-every 15 minutes
  Skin thermometer used to measure body temperature
Duration of operation | Perioperative period
  Duration of operation compared with the change in body temperature
Blood loss | Perioperative period
  Blood loss during the perioperative period
Shivering after the operation | Postoperative 1st hour every 10 minutes
  Assessment of shivering after operation in the recovery room with PAS score
Time to extubation | The end of the operation
  Time to extubation at the end of operation

CONTACTS AND LOCATIONS:
Overall Officials: Meral Kanbak, Prof, Study Chair — Hacettepe University; FİLİZ UZUMCUGIL, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University School of Medicine Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No